CLINICAL TRIAL: NCT04278820
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study of TQA3526 in the Treatment of Naive or Previously Treated PBC Patients
Brief Title: A Study of TQA3526 in the Treatment of Primary Biliary Cirrhosis (PBC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA3526-Ⅱ-01
Record Dates: First submitted 2020-01-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-12

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Climbing group (Experimental)
  Interventions: Drug: TQA3526; Drug: Placebo to match TQA3526
- Titration group (Experimental)
  Interventions: Drug: TQA3526; Drug: Placebo to match TQA3526
- Extension group (Experimental)
  Interventions: Drug: TQA3526; Drug: Placebo to match TQA3526

INTERVENTIONS:
Drug: TQA3526 — Tablet(s) administered orally once daily
Drug: Placebo to match TQA3526 — Tablet(s) administered orally once daily

SUMMARY:
TQA3526 is a modified bile acid and FXR agonist. FXR is a key regulator of bile acid synthesis and transport. Bile acids are used by the body to help with digestion. It is hypothesized that regular treatment with TQA3526 will improve liver function in persons with Primary Biliary Cirrhosis (PBC).

ELIGIBILITY:
Inclusion Criteria:

* 1.18 and 70 years old, male or female. 2.Proven as PBC, as demonstrated by the patient presenting with at least 2 of the following 3 diagnostic factors:

  * History of increased ALP levels for at least 3 months prior to Day 0 in previously treated PBC patients，or ALP levels increased during screening in treatment naive PBC patients； ② Positive AMA titer (>1:40 titer on immunofluorescence or M2 positive by ELISA) or PBC-specific antinuclear antibodies (anti-GP210 and anti-SP100 positive)； ③ Liver biopsy consistent with PBC within 24W prior to randomization； 3.ALP value between 1.67 and 10 × ULN; 4.Taking ursodeoxycholic acid (UDCA) for at least 12 months (stable dose for ≥ 3 months) prior to Day 0, or unable to tolerate UDCA (no UDCA for ≥ 3 months) prior to Day 0.

Exclusion Criteria:

* 1.Has other virus infected ; 2.History or presence of other concomitant liver diseases； 3.Presence of clinical complications of PBC or clinically significant hepatic decompensation； 4.Child-pugh grade B or C in patients with cirrhosis； 5.Creatinine (Cr) ≥1.5 times the upper limit of normal value and serum creatinine clearance rate <60mL/min； 6.ALT or AST>5×ULN；TBil>3×ULN； 7.Patients with a history of severe pruritus within 2 months prior to day 0; 8.History or presence of clinically concerning cardiac arrhythmias, the duration of the study may affect survival; 9.Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the intestine; 10.Medical conditions that may cause nonhepatic increases in ALP (e.g., Paget's disease) or which may diminish life expectancy to < 2 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Alkaline phosphatase (ALP) | Baseline up to 24w
  The reduction of ALP level from baseline to 24 weeks.

SECONDARY OUTCOMES:
Liver function：ALP (excluding 12W/24W), ALT, AST, GGT, TBA and Tbil | Baseline up to 2, 4, 8, 12, 14, 16, 20, 24 weeks
  The reduction of ALP , ALT, AST, GGT, TBA and Tbil from baseline to each time point.
Fasting lipid：LDL-C、HDL-C、TG and TC | Baseline up to 2, 4, 8, 12, 14, 16, 20, 24 weeks
  The rate of change of LDL-C、HDL-C、TG and TC from baseline to each time point.
Cmax | predose, Weeks 2, 4, 8, 12, 14, 16, 20, 24 : 0, 1.5, 3.5 hours following drug administration
  Maximum concentration of the analyte in plasma.
tmax | predose, Weeks 2, 4, 8, 12, 14, 16, 20, 24 : 0, 1.5, 3.5 hours following drug administration
  Time from dosing to maximum concentration
AUC0-∞ | predose, Weeks 2, 4, 8, 12, 14, 16, 20, 24 : 0, 1.5, 3.5 hours following drug administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
pharmacodynamics | Baseline up to 2, 4, 8, 12, 14, 16, 20, 24 weeks
  The rate of change of FGF-19、C4、IgG and IgM from baseline to each time point.
safety and tolerability: incidence of treatment emergent adverse events and serious treatment emergent adverse events | Baseline up to 2, 4, 8, 12, 14, 16, 20, 24 weeks
  Evaluate safety and tolerability as assessed by the incidence of treatment emergent adverse events and serious treatment emergent adverse events comparing TQA3526 to placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China